CLINICAL TRIAL: NCT05716191
Title: Study on the Relationship Between Iodine Nutrition and Thyroid Diseases in the Elderly
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tianjin Medical University (Other)
Collaborators: Tianjin Medical University General Hospital (Other); Shandong Provincial Institute for Endemic Disease Control (Unknown)
Responsible Party: Principal Investigator, Wenxing Guo, Lecturer, Tianjin Medical University
Other Study IDs: NSFC-82204041
Record Dates: First submitted 2022-12-21; First posted 2023-02-08 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Nutrition, Healthy; Elderly
Keywords: iodine; thyroid diseases; adults
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — 1.Urinary iodine concentration was measured by collecting spot urine and 24-h urine samples. 2.Blood samples were collected to evaluate thyroid function. 3.Thyroid B-ultrasonography was conducted to measure the thyroid volume and thyroid nodule. 4.Saliva samples were collected to measure saliva iodine. 5.The iodine dietary frequency questionnaire was used to assess the long-term iodine intake level of the subjects.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Naturally different iodine levels exposure — A cross-sectional survey of thyroid disease in elderly people in areas with different iodine nutrition backgrounds

SUMMARY:
The aging trend of China's population is intensifying. More than 50% of the elderly in China suffer from thyroid disease. Thyroid dysfunction in the elderly increases the risk of cardiovascular and metabolic diseases. Even if thyroid-stimulating hormone (TSH) is within the normal range, brain atrophy and infarction-like vascular damage in elderly males will be aggravated with the increased TSH level. Iodine is an essential component of thyroid hormones. Iodine deficiency or excess may lead to a series of thyroid diseases. The risk threshold of iodine intake in the elderly is unknown. The goal of this observational study is to clarify the relationship between thyroid diseases and iodine intake in the elderly. The aims are:

1. to clarify the differences in the prevalence of thyroid diseases in the elderly with different iodine nutrition backgrounds.
2. to analyze the effects of mild iodine deficiency and iodine excess on the thyroid health of the elderly.
3. to explore the hazard threshold of iodine intake for old people.
4. to compare the differences in thyroid disease and iodine nutritional status between young and middle-aged people and old people.

DETAILED DESCRIPTION:
Part 1：A cross-sectional survey of thyroid diseases in adults in different iodine nutrition background areas.

Investigators will separately include adults ( middle-aged people and old people) in iodine-deficient, iodine-appropriate, and iodine-excessive areas. Venous blood will be collected to measure thyroid function and serum iodine. Thyroid volume and nodular disease were determined by B-ultrasonography. Drinking water, saliva and 24-h and spot urinary samples will be collected to precisely evaluate the daily iodine intake. Multiple indicators were used to accurately evaluate the iodine intake level of the subjects, and understand the differences in the prevalence of thyroid diseases in the elderly under different iodine nutrition backgrounds. Besides, the differences in thyroid disease and iodine nutritional status between young and middle-aged people and old people will be compared.

Part 2：A survey on the iodine nutrition status in the elderly with/without thyroid disease in iodine-appropriate areas.

Investigators will collect basic information (height, weight, age, other medical histories, etc.) and thyroid disease history information. Thyroid B-ultrasound and thyroid function tests were used to understand the current thyroid status of the elderly. The iodine dietary frequency questionnaire was used to assess the long-term iodine intake level of the survey subjects, and spot urinary iodine, 24-h urinary iodine and salivary iodine were used to assess the short-term iodine intake level of the survey subjects.

ELIGIBILITY:
Inclusion Criteria:

1. adults with at least 5 years of local residence;

Exclusion Criteria:

1. adults with family genetic diseases
2. adults with special dietary habits
3. adults taking iodine-containing drugs or supplements
4. adults with protein or nutritional deficiencies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Elderly people with different levels of iodine exposure.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-02-17 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
thyroid function Indicators | 2 years
  Blood samples were collected to evaluate thyroid function.
thyroid volume | 2 years
  Thyroid volume was measured by B-ultrasound.
thyroid nodules | 2 years
  thyroid nodules were measured by B-ultrasound.
concentration of urinary iodine | 2 years
  The midstream urine samples were collected.
concentration of salivary iodine | 2 years
  The salivary samples were collected.
dietary iodine intake | 2 years
  Dietary iodine was measured by idine dietary frequency questionnaire.

SECONDARY OUTCOMES:
free triiodothyronine (FT3) | 2 years
  thyroid function Indicators
free thyroxine (FT4) | 2 years
  thyroid function Indicators
thyroid-stimulating hormone (TSH) | 2 years
  thyroid function Indicators
thyroperoxidase antibody (TPOAb) | 2 years
  thyroid function Indicators
thyroglobulin antibody (TGAb) | 2 years
  thyroid function Indicators

CONTACTS AND LOCATIONS:
Overall Officials: Wenxing Guo, Doctor, Study Chair — Public Health School, Tianjin Medical University
Locations (3):
- China (3):
  - Gansu provincial center for disease control and prevention, Lanzhou, Gansu
  - Shandong provincial institute for endemic disease control, Jinan, Shandong
  - Tianjin Medical University, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: Undecided
The data of the study are available from the project leader upon reasonable request.

REFERENCES:
- [Background] Zimmermann MB, Boelaert K. Iodine deficiency and thyroid disorders. Lancet Diabetes Endocrinol. 2015 Apr;3(4):286-95. doi: 10.1016/S2213-8587(14)70225-6. Epub 2015 Jan 13. PMID 25591468
- [Background] Leung AM, Braverman LE. Consequences of excess iodine. Nat Rev Endocrinol. 2014 Mar;10(3):136-42. doi: 10.1038/nrendo.2013.251. Epub 2013 Dec 17. PMID 24342882
- [Background] Li Y, Teng D, Ba J, Chen B, Du J, He L, Lai X, Teng X, Shi X, Li Y, Chi H, Liao E, Liu C, Liu L, Qin G, Qin Y, Quan H, Shi B, Sun H, Tang X, Tong N, Wang G, Zhang JA, Wang Y, Xue Y, Yan L, Yang J, Yang L, Yao Y, Ye Z, Zhang Q, Zhang L, Zhu J, Zhu M, Ning G, Mu Y, Zhao J, Shan Z, Teng W. Efficacy and Safety of Long-Term Universal Salt Iodization on Thyroid Disorders: Epidemiological Evidence from 31 Provinces of Mainland China. Thyroid. 2020 Apr;30(4):568-579. doi: 10.1089/thy.2019.0067. Epub 2020 Mar 24. PMID 32075540
- [Background] Miller JC, MacDonell SO, Gray AR, Reid MR, Barr DJ, Thomson CD, Houghton LA. Iodine Status of New Zealand Elderly Residents in Long-Term Residential Care. Nutrients. 2016 Jul 23;8(8):445. doi: 10.3390/nu8080445. PMID 27455319
- [Background] Laurberg P, Cerqueira C, Ovesen L, Rasmussen LB, Perrild H, Andersen S, Pedersen IB, Carle A. Iodine intake as a determinant of thyroid disorders in populations. Best Pract Res Clin Endocrinol Metab. 2010 Feb;24(1):13-27. doi: 10.1016/j.beem.2009.08.013. PMID 20172467
- [Background] Limanova Z. [Thyroid disease in the elderly]. Vnitr Lek. 2018 Winter;64(11):993-1002. Czech. PMID 30606015
- [Background] Zhai X, Zhang L, Chen L, Lian X, Liu C, Shi B, Shi L, Tong N, Wang S, Weng J, Zhao J, Teng X, Yu X, Lai Y, Wang W, Li C, Mao J, Li Y, Fan C, Li L, Shan Z, Teng W. An Age-Specific Serum Thyrotropin Reference Range for the Diagnosis of Thyroid Diseases in Older Adults: A Cross-Sectional Survey in China. Thyroid. 2018 Dec;28(12):1571-1579. doi: 10.1089/thy.2017.0715. Epub 2018 Nov 27. PMID 30351201
- [Background] Barbesino G. Thyroid Function Changes in the Elderly and Their Relationship to Cardiovascular Health: A Mini-Review. Gerontology. 2019;65(1):1-8. doi: 10.1159/000490911. Epub 2018 Jul 20. PMID 30032140
- [Background] Iacone R, Iaccarino Idelson P, Russo O, Donfrancesco C, Krogh V, Sieri S, Macchia PE, Formisano P, Lo Noce C, Palmieri L, Galeone D, Rendina D, Galletti F, Di Lenarda A, Giampaoli S, Strazzullo P, On Behalf Of The Minisal-Gircsi Study Group. Iodine Intake from Food and Iodized Salt as Related to Dietary Salt Consumption in the Italian Adult General Population. Nutrients. 2021 Sep 30;13(10):3486. doi: 10.3390/nu13103486. PMID 34684487
- [Derived] Jin Q, Wang Z, Li J, Zhang H, Liu M, Wang C, Guo W, Zhang W. Iodine Excess Is Associated with Thyroid Dysfunction Among the Elderly. Biol Trace Elem Res. 2025 Jul;203(7):3470-3478. doi: 10.1007/s12011-024-04420-0. Epub 2024 Oct 23. PMID 39441230